CLINICAL TRIAL: NCT03073954
Title: The Feasibility of Working Memory Training in COPD Patients and the Efficacy on Cognitive Performance, Self-Control and Stress Response
Brief Title: Working Memory Training in COPD Patients: the Cogtrain-Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Eatwell (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NL59883.068.17
Record Dates: First submitted 2017-01-31; First posted 2017-03-08 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2018-03

CONDITIONS: COPD; Cognitive Impairment
Keywords: Health Behavior; Executive function; Working-memory training; Feasibility; Impulsivity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction; Health Behavior; Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working memory training (Active Comparator): Working memory training that increases with difficulty if participants answer two subsequent questions correctly, and standardised healthy lifestyle coaching.
  Interventions: Other: Working memory training; Behavioral: Standardised healthy lifestyle coaching
- Sham working memory training (Sham Comparator): Working memory training that does not increase in difficulty, and standardised healthy lifestyle coaching.
  Interventions: Other: Working memory training; Behavioral: Standardised healthy lifestyle coaching

INTERVENTIONS:
Other: Working memory training — The working memory intervention training programme consists of a domain-general cognitive working memory training programme. One training session will take 20 to 30 minutes, and participants will have to complete approximately 40 cognitive training sessions.
  The sham treatment is the same as the intervention training however it does not increase in difficulty. Participants are presented with the same task at the same level of difficulty over and over again. Thus a training effect is not expected.
Behavioral: Standardised healthy lifestyle coaching — Participants will receive standardised healthy living coaching focusing on healthy diet and daily physical activity.

SUMMARY:
General cognitive impairment is highly prevalent in chronic obstructive pulmonary disease (COPD) patients. Domain-specific cognitive impairments include deficits in domains such as cognitive flexibility, verbal memory, working memory, planning, and psychomotor speed; which in general are associated with poor health behaviours, such as infrequent exercising and poor diet. Additional cognitive training may reverse these effects. Recent evidence suggests that working memory training is linked to self-control and, indirectly, to improved lifestyle behaviour including increased physical activity. The investigators hypothesise that enhancing cognitive performance through administering specific working memory training not only improves cognitive function but that it facilitates better adherence to a more active lifestyle and a healthier diet in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of COPD based on the Global Initiative for Chronic obstructive Lung Disease (GOLD) guidelines
* Patients also need to provide written informed consent
* Be motivated as evaluated by the self-determination questionnaire

Exclusion Criteria:

* Disease and or disability limiting the ability to undergo a neuropsychological testing battery and/or to follow a working memory training (e.g., blindness)
* Neurological disorders (e.g., Alzheimer's Disease or cerebrovascular disease)
* Insufficient mastery of the Dutch language
* Individuals who during the study period are or will be participating in a PR programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the cognitive training in COPD patients as measured through training compliance. | 6 months
  The compliance as well as the acceptability of working memory training in the COPD patient population will be investigated
Change in cognitive performance before and after working memory training as assessed through a cognitive test performance battery. | 6 months
  Improvement in cognitive flexibility, planning, and working memory.

SECONDARY OUTCOMES:
Self-control (impulsivity) | 6 months
  This will be measured using the stop signal task.
Chronic stress levels as measured through hair levels of cortisol | 6 months
  An objective measure of stress levels experienced over the last 3 months will be measured using cortisol extracted from a hair sample.
Stress levels as measured through the salivary cortisol awakening response | 6 months
  An objective measure of stress will be measured using salivary cortisol awakening response
Stress perception as assessed through a perceived stress scale. | 6 months
  A subjective measure of chronic stress will be measured using the perceived stress scale score.
Acute stress as assessed through the socially evaluated cold pressor test | 6 months
  Acute stress will be measured using the socially evaluated cold pressor test, heart rate is also monitored.
Daily physical activity level | 6 months
  Physical activity data will be collected by an accelerometer using step counts.
Mental health, depressive symptoms assessed via the BDI-II | 6 months
  Mental health with respect to depression will be evaluated using the Beck Depression Inventory-second edition (BDI-II)
Mental health, anxiety symptoms assessed via the GAD-7 | 6 months
  Mental health with respect to anxiety will be evaluated using the Generalised Anxiety Disorder 7 (GAD-7)
Physical performance assessed through the 6 minute walk test | 6 months
  Changes in physical performance will be assessed using the 6-minute walking test (6MWT).Two six-minute walk tests (6MWT) will be performed according to ERS/ATS guidelines to measure functional exercise capacity. The best 6MWT will be expressed in percentage of predicted values.
Self-determination questionnaire | 6 months
  Motivation will be prior to the enrolment of participants in this study in order to include patients who are motivated to initiate and continue our working memory training. The self-made questionnaire evaluates patient's reasons for participating in the study in order to assess their intrinsic motivation.
Short Performance Battery | 6 months
  The SPPB consists of three types of physical manoeuvres: the balance tests, the gait speed test, and the chair stand test. The results of the different tests result in a score which will be used for analysis.
Changes in dietary intake over the intervention period | 6 months
  Changes in dietary intake over the intervention period will be assessed using a food frequency questionnaire.
Medication adherence | 6 months
  Medication adherence will be measured using a sem
Regulation of Eating Behavior Scale (REBS) | 6 months
  Changes in eating behavior motivation will be investigated using the REBS.
Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) Regulation | 6 months
  Changes in exercise motivation will be investigated using the BREQ-2
COPD Assessment test (CAT) | 6 months
  Impact of the intervention on quality of life will be done using the brief CAT questionnaire.
Anthropometry | 6 months
  Alterations in Anthropometical measures will be evaluated using waist circumference, biometric impedance, and body weight (BMI).
Manipulation Check | 6 months
  Participants will be asked to recall key health messages from their personalized healthy lifestyle advice sessions. Responses will be scored as follows: 0 points - field blank or no recall of the message content; 1 point - key points not directly related to the message themes; 2 points - key points directly related to the message themes.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No